CLINICAL TRIAL: NCT02841397
Title: Validation of a Pulse Oximetry Based Hemoglobin Measurement System. Comparison of Plethysmographic Variability Index to Standard Methods of Guiding Fluid and Transfusion Management in the Critically Ill Adult Patients. Validation of Clinical Efficacy of ORI for Supplemental Oxygen Titration
Brief Title: Validation of Noninvasive Hemoglobin, Comparison of PVI to Standard Methods, and Validation of Clinical Efficacy of ORI
Status: Completed | Type: Interventional
Sponsor: Masimo Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: DORO0001
Record Dates: First submitted 2016-07-13; First posted 2016-07-22 (Estimated); Results first posted 2021-10-21 (Actual); Last update posted 2021-10-21 (Actual); Status verified 2021-09

CONDITIONS: Surgery

STUDY DESIGN:
Oversight: Unapproved Device: Yes

ARMS (1):
- Test group (Experimental): All subjects will be enrolled into the test group and will receive Masimo Pulse CO-Oximeter for measurement of various physiological parameters.
  Interventions: Device: Masimo Pulse CO-Oximeter

INTERVENTIONS:
Device: Masimo Pulse CO-Oximeter — Noninvasive pulse oximeter with various features for measurement of hemoglobin, pleth variability index, and oxygen reserve index

SUMMARY:
The study goal is to establish the correlation of hemoglobin values determined by the noninvasive pulse oximetry-determined hemoglobin (SpHb) system with hemoglobin as measured by other validated devices. The study will also evaluation oxygen reserve index (ORI) to correlate with partial pressure of oxygen (PaO2), and to evaluate pleth variability index (PVI) with stroke volume variation (SVV) or pulse pressure variation (PPV) values.

ELIGIBILITY:
Inclusion Criteria:

* Admitted into the ICU
* Aged 18 years or older
* Mechanically ventilated
* Arterial line placed
* Vigileo/Flotrac System being used for guidance of fluid management

Exclusion Criteria:

* Pregnancy
* Prisoner status
* Extreme hemodynamic instability
* Multiple vasopressors in use with questionable peripheral blood flow
* Lack of appropriate sites for sensor placement
* Patient or patient's legal representative refusal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-03-09 (Actual); Primary Completion 2017-10-11 (Actual); Study Completion 2017-10-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Loma Linda University Medical Center, Loma Linda, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Test Group
Started | 50
Completed | 48
Not Completed | 2

BASELINE CHARACTERISTICS:
Arm/Group | Test Group
Number analyzed (Participants) | 50
Age, Categorical [Count of Participants; unit: Participants] — Population: There were four subjects that did not complete the study.
  Participants
    number analyzed (Participants) | 48
    <=18 years | 1
    Between 18 and 65 years | 30
    >=65 years | 17
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Please see reasons provided above.
  Participants
    number analyzed (Participants) | 48
    Female | 26
    Male | 22
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants] — Population: Please see reasoning above.
  participants
    United States: number analyzed (Participants) | 48
    United States | 48

OUTCOME MEASURES:

1. Primary Outcome: Noninvasive Pulse Oximetry-determined SpHb Bias
Description: Accuracy of SpHb will be determined by comparing it to the hemoglobin value obtained from a reference blood sample and calculating the accuracy root mean square (Arms) error value. In order to obtain the Arms value, the blood sample hemoglobin value is subtracted from SpHb value for a number of samples, the average of this difference is computed as the bias. The standard deviation of the differences is computed as the precision. The square root of the sum of the squares of bias and precision is computed as the Arms Error value.
Time Frame: Duration of study participation is up to three days.
Population: A total of 12 subjects were excluded from data analysis Subjects were excluded from data analysis for different reasons. Reason 1: Blood sample could not be analyzed because received out of analyzer required time window Reason 2: Sensor data is not available Reason 3: No time matched sensor and blood sample data pair for analysis Reason 4: Reference tHb error. tHb difference >1g/dL between different methods
Measure: Number; unit: g/dL
Arm/Group | Test Group
Number analyzed (Participants) | 34
g/dL | 0.9

2. Primary Outcome: Correlation of PVI Measurement Compared With PPV or SVV
Description: Correlation of PVI measurement compared with pulse pressure variation PPV or stroke volume variation (SVV) measurement from arterial catheter
Time Frame: Duration of study participation is up to three days.
Population: There was no reference SVV or PPV data available for PVI data analysis.
Arm/Group | Test Group
Number analyzed (Participants) | 0

3. Primary Outcome: Correlation of "ORI" With Partial Pressure of Oxygen (PaO2) "PaO2" Measurement From Blood Gas Analysis
Description: Concordance will be determined by comparing the trending ability of the Oxygen Reserve Index (ORI) measurement of the sensor with that of Partial Pressure of Oxygen in Blood (PaO2).
Time Frame: Duration of study participation is up to three days.
Population: Data from 8 subjects were obtained. At least two samples per subject are required to compare ORI trending ability; however, only 1 sample was obtained from each subject which precluded conduct of any data analysis.
Arm/Group | Test Group
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse events were monitored throughout study duration, which was up to three days.
Arm/Group | Test Group
All-Cause Mortality (participants affected / at risk) | 0/50
Serious Adverse Events (participants affected / at risk) | 0/50
Other Adverse Events (participants affected / at risk) | 0/50

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-08-10): https://cdn.clinicaltrials.gov/large-docs/97/NCT02841397/Prot_SAP_000.pdf